CLINICAL TRIAL: NCT07170215
Title: Effect of Anti-gravity Treadmill Training After Total Hip Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rijeka (Other)
Responsible Party: Principal Investigator, Mirela Vuckovic, Assist. prof, University of Rijeka
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: THR-2025
Record Dates: First submitted 2025-09-05; First posted 2025-09-12 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Osteoarthritis, Hip
Keywords: pain; functional mobility; muscle strenght; total hip arthroplasty; THA
MeSH Terms: conditions — Osteoarthritis, Hip; Pain

STUDY DESIGN:
Intervention Model Description: Patients were randomly assigned to one of two groups: the experimental group (EG) (n = 18) received antigravity treadmill therapy in combination with a standard rehabilita-tion protocol and the control group (CG) (n = 16) followed only the conventional rehabili-tation protocol.
Masking Description: Masking was not possible.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (EG) (Experimental): Each session included 25 minutes of individualized therapeutic exercises focused on bre-athing, mobility, strength, and balance. In addition, participants received 25 minutes of electrical stimulation of the quadriceps femoris muscle and 25 minutes of hydrotherapy in a swimming pool, for a total of 75 minutes of therapy per session. The experimental group (EG) also completed 20 minutes of daily exercise on an antigravity treadmill (ALTERG VIA, Lifeward CA, Inc., Milmont Drive, Fremont, CA, USA), supervised by a physiothera-pist
  Interventions: Device: antigravity treadmill (ALTERG VIA, Lifeward CA, Inc., Milmont Drive, Fremont, CA, U-SA)
- control group (CG) (No Intervention): Each session inclu-ded 25 minutes of individualized therapeutic exercises focused on breathing, mobility, strength, and balance. In addition, participants received 25 minutes of electrical stimula-tion of the quadriceps femoris muscle and 25 minutes of hydrotherapy in a swimming pool, for a total of 75 minutes of therapy per session.

INTERVENTIONS:
Device: antigravity treadmill (ALTERG VIA, Lifeward CA, Inc., Milmont Drive, Fremont, CA, U-SA) — Antigravity treadmill training in the experimental group (EG) involved walking in a straight line at a self-selected, com-fortable pace-without running, shortness of breath, or pain. The treadmill's chamber was set to reduce the participant's effective body weight to 20% of their actual body weight (slight unloading was applied to reduce the need for handrail support and to prevent the use of compensatory mechanisms).
  Arms: experimental group (EG)

SUMMARY:
Background/Objectives: Total hip arthroplasty is one of the most common orthopedic procedures. When the surgery is successful and followed by high-quality physiotherapy, patients' quality of life usually improves and they return to their daily activities more qui-ckly.. Rehabilitation methods and medical devices are constantly evolving, to accelerate functional improvement. The aim of the study is to investigate the impact of the antigra-vity treadmill on the functional outcomes after total hip arthroplasty. Methods: A single centre, randomised, controlled, open label trial was conduct in Hospital for Medical Re-habilitation of the Heart and Lung Diseases and Rheumatism Thalassotherapia Opatija. 34 subjects were randomly divided into two groups: experimental (18) and control (16). The outcome measures included strength of the abductor muscles, range of motion, visual analogue scale, and Timed Up and Go test and 40-meter Fast Paced Walk test.

ELIGIBILITY:
Inclusion Criteria:

* The inclusion criteria was primary osteoarthritis of the hip joint.

Exclusion Criteria:

* Exclusion criteria included: Undergoing surgery using a different technique, revision hip replacement, acute illness, cognitive impairment, and declining participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2023-01-15 (Actual); Primary Completion 2023-07-30 (Actual); Study Completion 2023-07-30 (Actual)

PRIMARY OUTCOMES:
hip abductor muscle strength | From enrollment to the end of treatment was 3 weeks.
  The effects of the antigravity treadmill on hip abductor muscle strength was the primary outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Thalassotherapia Opatija, Rijeka, Croatia

IPD SHARING:
Plan to Share IPD: No